CLINICAL TRIAL: NCT00958191
Title: An Open-label, Prospective, Post-market, Historically Controlled, Multi-center Clinical Evaluation of the Trident® X3 Polyethylene Acetabular Inserts.
Brief Title: Trident® X3 Polyethylene Insert Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 57
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trident® X3 Polyethylene Insert (Other): Participants who received the Trident® X3 Polyethylene Insert.
  Interventions: Device: Trident® X3 Polyethylene Insert

INTERVENTIONS:
Device: Trident® X3 Polyethylene Insert — Trident® X3 Polyethylene Insert

SUMMARY:
The primary objective of the study is to demonstrate the linear wear rates of the Trident® X3 polyethylene insert are superior to a polyethylene control group wear rate at 5 years postoperative. This measurement will be evaluated by comparing digitized images of serial radiographs obtained over a follow-up period of 5-years.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, historical-controlled clinical evaluation of the Trident® X3 Polyethylene insert. The device is commercially available in the United States where the study is being conducted. The study device, the Stryker Orthopaedics Trident® X3 polyethylene insert, is used for the replacement of the bearing surface of the acetabulum to relieve pain, instability, and the restriction of motion due to degenerative bone disease, including osteoarthritis, rheumatoid arthritis, trauma, or failure of other devices. The control device, the Stryker Orthopaedics N2VAC polyethylene insert, is also used for the replacement of the bearing surface of the acetabulum to relieve pain, instability, and the restriction of motion due to degenerative bone disease, including osteoarthritis, rheumatoid arthritis, trauma, or failure of other devices.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed an IRB-approved, study specific Patient Informed Consent Form.
2. The patient is a candidate for a primary total hip replacement with cementless acetabular and femoral components.
3. The patient has a primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD). Patient must have diagnosis of osteoarthritis (OA), traumatic arthritis (TA), avascular necrosis (AVN), slipped capital epiphysis, pelvic fracture, femoral fracture, failed fracture fixation, or diastrophic variant.
4. The patient is a male or non-pregnant female patient ages 21 to 75.
5. The patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. The patient has an active infection with the affected hip joint.
2. The patient requires revision surgery of a previously implanted total hip arthroplasty or hip fusion to the affected joint.
3. The patient has a BMI >45.
4. The patient has a neuromuscular or neurosensory deficiency, which limits ability to evaluate the safety and efficacy of the device.
5. The patient has diagnosed systemic disease (i.e. Paget's disease, renal osteodystrophy).
6. The patient is immunologically suppressed or receiving chronic steroids in excess of 5mg per day.
7. The patient has a recent history of substance dependency that may result in deviations from the evaluation schedule.
8. The patient is a prisoner.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-05; Primary Completion 2012-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D'Antonio, MD, Study Chair — Greater Pittsburgh Orthopaedic Association; Benjamin Bierbaum, MD, Principal Investigator — New England Baptist Hospital Deptartment of Orthopaedics; Peter Bonutti, MD, Principal Investigator — Bonutti Clinic; William Capello, MD, Principal Investigator — Indiana University School of Medicine; Michael Taunton, MD, Principal Investigator — Mayo Clinic Department of Orthopaedic Surgery; Robert Johnson, MD, Principal Investigator — University of Vermont College of Medicine Department of Orthopaedics & Rehabilitation; J. Wesley Mesko, MD, Principal Investigator — Michigan Orthopaedic Center; James R Roberson, MD, Principal Investigator — Emory Orthopaedics; John Wright, MD, Principal Investigator — New West Orthopaedics; Daniel Ward, MD, Principal Investigator — New England Baptist Hospital Department of Orthopaedics; Russell Meldrum, MD, Principal Investigator — Indiana University School of Medicine; J. Andrew Parr, MD, Principal Investigator — Indiana University School of Medicine; Steven Incavo, MD, Principal Investigator — University of Vermont; Greg Erens, MD, Principal Investigator — Emory Orthopaedics; Robert Trousdale, MD, Principal Investigator — Mayo Clinic Department of Orthopaedic Surgery; Alren Hanssen, MD, Principal Investigator — Mayo Clinic Department of Orthopaedic Surgery
Locations (9):
- United States (9):
  - Emory University, Atlanta, Georgia
  - Bonutti Research Inc., Effingham, Illinois
  - Indiana University, Indianapolis, Indiana
  - New England Baptist Hospital, Boston, Massachusetts
  - J. Wesley Mesko, MD, Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Good Samaritan Hospital, Kearney, Nebraska
  - Greater Pittsburgh Orthopaedics Assoc, Pittsburgh, Pennsylvania
  - University of Vermont College of Medicine, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For bilateral hip replacement participants, if one hip completed primary endpoint #1 the participant is counted as completed. If one hip was censored, but the other hip was not, the hip is counted as censored, but the participant is not.
Pre-assignment Details: 250 participants/271 hips enrolled - 29 participants/31 hips censored= 221 participants/240 hips followed. There were 5 revisions, but one bilateral participant had one hip revised and the other hip completed the primary endpoint. This participant is counted as completed and not in the revision category.
Units Other Than Participants: hips
Groups:
- Trident® X3 Polyethylene Insert: Participants who received the Trident X3 polyetheylene insert can have one or both hips replaced. If both hips were replaced, but one hip completed the primary endpoint, the participant is counted as completed.
Period: Overall Study
Arm/Group | Trident® X3 Polyethylene Insert
Started | 221; 240 hips
Completed (Complete/Not completed counts are based on participant status at the 5 yr primary outcome interval.) | 110; 118 hips
Not Completed | 111; 122 hips
Not completed — Death | 4
Not completed — Lost to Follow-up | 5
Not completed — Inadequate 5 yr x-ray quality | 10
Not completed — Unable/Unwilling to Return/Withdrawal | 21
Not completed — Revision of study device | 4
Not completed — Site termination | 11
Not completed — No 5 yr x-rays | 56

BASELINE CHARACTERISTICS:
Population: Includes participants who received the Trident X3 polyetheylene insert and were not censored from analysis.
Groups:
- Trident® X3 Polyethylene Insert: All subjects who recieved the Trident X3 insert.
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 221
Age, Continuous [Mean (Standard Deviation); unit: years] — For bilateral participants, age at the time of surgery for the first hip enrolled is used for the baseline measurement.
  years | 62.04 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 105
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 221

OUTCOME MEASURES:

1. Primary Outcome: Mean Linear Wear Rate at 5 Years
Description: Linear wear rates are defined as the annual rate of removal of the polyethylene from the polyethylene insert determined by comparing digitized images of serial radiographs obtained over the follow-up period of 5 years
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mm/year
Units Other Than Participants: Hips
Groups:
- Trident® X3 Polyethylene Insert: Participants who received theTrident® X3 Polyethylene Insert
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 110
Number analyzed (Hips) | 118
mm/year | 0.016 (0.068)

2. Primary Outcome: Rate of Incidence of Revision of Component for Any Reason
Description: Revision of any component is defined as surgical removal and replacement of the femoral component, acetabular shell, acetabular insert and/or femoral head.
Time Frame: 5 year
Population: Difference of 5 participants from the participant flow completed (=110): 4 participants are included in the revision category of the participant flow and one participant had revision of only the femoral head & stem but later withdrew from the study & is included in the withdrawal category of the participant flow.
Measure: Number; unit: percentage of hips undergoing revision
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 115
Number analyzed (Hips) | 124
percentage of hips undergoing revision | 4.84

3. Secondary Outcome: Linear Wear Rate of the Trident X3 Polyethylene Insert
Description: Linear wear rates are defined as the annual rate of removal of the polyethylene from the polyethylene insert determined by comparing digitized images of serial radiographs obtained over the follow-up period.
  NOTE: 2 year linear and volumetric wear was not calculated for the following reason: To determine polyethylene wear, the total femoral head penetration is first calculated from the radiographs.The femoral head penetration has two components namely wear and creep (or bedding-in). It is not possible to separate the total penetration in to two components. The creep of the polyethylene starts from the date of surgery and continues up to 12-24 months. Therefore, the head penetration value at 2-years is dominated by Creep rather than wear.
Time Frame: 2, 3 and 4 year films collected; 3 and 4 year wear assessed
Population: Participants/hips with available data. Overall number of participants and units analyzed is based upon the 3 year population.
Measure: Mean (Standard Deviation); unit: mm/year
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 140
Number analyzed (Hips) | 149
mm/year
  3 year mean wear rate | 0.022 (0.133)
  4 year mean wear rate: number analyzed (Participants) | 127
  4 year mean wear rate: number analyzed (Hips) | 134
  4 year mean wear rate | 0.024 (0.087)

4. Secondary Outcome: Volumetric Wear Rate of the Trident X3 Polyethylene Insert
Description: Volumetric wear rate is calculated using a formula based on the cylindrical wear pattern perpendicular to the face of the cup and the mean linear wear rate.
  NOTE: 2 year linear and volumetric wear was not calculated for the following reason: To determine polyethylene wear, the total femoral head penetration is first calculated from the radiographs.The femoral head penetration has two components namely wear and creep (or bedding-in). It is not possible to separate the total penetration in to two components. The creep of the polyethylene starts from the date of surgery and continues up to 12-24 months. Therefore, the head penetration value at 2-years is dominated by Creep rather than wear.
Time Frame: 2, 3, 4 and 5 year films collected; 3, 4 and 5 year wear assessed
Population: as for outcome 3
Measure: Number; unit: cubic mm/year
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 140
Number analyzed (Hips) | 149
cubic mm/year
  3 year volumetric wear rate | 17.9
  4 year volumetric wear rate: number analyzed (Participants) | 127
  4 year volumetric wear rate: number analyzed (Hips) | 134
  4 year volumetric wear rate | 19.1
  5 year volumetric wear rate: number analyzed (Participants) | 110
  5 year volumetric wear rate: number analyzed (Hips) | 118
  5 year volumetric wear rate | 13.3

5. Secondary Outcome: Radiographic Stability
Description: Radiographic stability is defined as having all of the following: no radiographic indication of progressive radiolucent lines greater than or equal to 2 mm around the entire acetabular cup, no radiographic indication of acetabular cup migration of greater than or equal to 3 mm, no radiographic indication of progressive radiolucent lines greater than or equal to 2 mm around the entire femoral component, and no radiographic indication of progressive subsidence of the femoral component of greater than or equal to 5 mm. Radiographs are evaluated at 1,2,3,4 and 5 years.
Time Frame: 1,2,3,4 and 5 years
Population: Participants/hips with available data. Overall number of participants and units analyzed is based upon the 1 year population.
Measure: Number; unit: hips evaluated as unstable on radiograph
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 197
Number analyzed (Hips) | 214
hips evaluated as unstable on radiograph
  Radiographically unstable at 1 year | 0
  Radiographically unstable at 2 years: number analyzed (Participants) | 179
  Radiographically unstable at 2 years: number analyzed (Hips) | 195
  Radiographically unstable at 2 years | 0
  Radiographically unstable at 3 years: number analyzed (Participants) | 155
  Radiographically unstable at 3 years: number analyzed (Hips) | 166
  Radiographically unstable at 3 years | 0
  Radiographically unstable at 4 years: number analyzed (Participants) | 142
  Radiographically unstable at 4 years: number analyzed (Hips) | 153
  Radiographically unstable at 4 years | 0
  Radiographically unstable at 5 years: number analyzed (Participants) | 129
  Radiographically unstable at 5 years: number analyzed (Hips) | 138
  Radiographically unstable at 5 years | 0

6. Secondary Outcome: Mean Harris Hip Score (HHS) to Assess Change
Description: The change in HHS is reported by comparing the mean preoperative, 1, 3 and 5 year postoperative scores that assess pain, function, joint deformity and range of motion. Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score less than or equal to 79 is considered fair-poor.
  90 - 100 = excellent
  80 - 89 = good
  70 - 79 = fair
  0 - 69 = poor
Time Frame: pre-operative, 1,3 and 5 years
Population: Participants/hips with available data. Overall number of participants and units analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 217
Number analyzed (Hips) | 236
units on a scale
  HHS Mean Preoperative Score | 53.01 (13.68)
  HHS Mean 1 Year Score: number analyzed (Participants) | 194
  HHS Mean 1 Year Score: number analyzed (Hips) | 211
  HHS Mean 1 Year Score | 94.41 (8.75)
  HHS Mean 3 Year Score: number analyzed (Participants) | 147
  HHS Mean 3 Year Score: number analyzed (Hips) | 158
  HHS Mean 3 Year Score | 95.32 (8.32)
  HHS Mean 5 year Score: number analyzed (Participants) | 114
  HHS Mean 5 year Score: number analyzed (Hips) | 121
  HHS Mean 5 year Score | 94.05 (8.70)
Statistical Analysis 1: Comparison: Trident® X3 Polyethylene Insert; Change in HHS from pre-op to 1 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 2: Comparison: Trident® X3 Polyethylene Insert; Change in HHS from pre-op to 3 years; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 3: Comparison: Trident® X3 Polyethylene Insert; Change in HHS from pre-op to 5 years; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

7. Secondary Outcome: Mean Harris Hip Score (HHS) Pain Score to Assess Change
Description: The change in HHS Pain is reported by comparing the mean preoperative, 1, 3 and 5 year postoperative pain scores. Scores can range from 0 to 44, with 0 indicating totally disabling pain and 44 indicating no pain or pain that is ignored.
  * None or ignores it = 44 points
  * Slight, occasional, no compromise in activities = 40 points
  * Mild pain, no effect on average activities, rarely moderate pain with unusual activity;may take aspirin = 30 points
  * Moderate pain, tolerable, but makes concessions to pain. Some limitation of ordinary activity or work. May require occasional pain medication stronger than aspirin = 20 points
  * Marked pain, serious limitation of activites = 10 points
  * Totally disabled, crippled, pain in bed, bedridden = 0 points
Time Frame: pre-operative, 1,3, and 5 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 221
Number analyzed (Hips) | 240
units on a scale
  HHS Pain Mean Preoperative Score | 16.73 (8.24)
  HHS Pain Mean 1 Year Score: number analyzed (Participants) | 200
  HHS Pain Mean 1 Year Score: number analyzed (Hips) | 217
  HHS Pain Mean 1 Year Score | 41.52 (5.64)
  HHS Pain Mean 3 Year Score: number analyzed (Participants) | 156
  HHS Pain Mean 3 Year Score: number analyzed (Hips) | 168
  HHS Pain Mean 3 Year Score | 42.50 (4.89)
  HHS Pain Mean 5 Year Score: number analyzed (Participants) | 123
  HHS Pain Mean 5 Year Score: number analyzed (Hips) | 130
  HHS Pain Mean 5 Year Score | 41.75 (5.99)
Statistical Analysis 1: Comparison: Trident® X3 Polyethylene Insert; Change in Harris Hip Pain Score from pre-op to 1 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 2: Comparison: Trident® X3 Polyethylene Insert; Change in Harris Hip Pain Score from pre-op to 3 years; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 3: Comparison: Trident® X3 Polyethylene Insert; Change in Harris Hip Pain Score from pre-op to 5 years; Test type: Superiority or Other; p < 0.0001, Sign test

8. Secondary Outcome: Mean Harris Hip Score (HHS) Range of Motion (ROM) Score to Assess Change
Description: The change in HHS ROM is reported by comparing the mean preoperative, 1, 3 and 5 year postoperative scores. Scores can range from 0 (worst) to 5 (best). The degrees of motion are measured for hip flexion, abduction, adduction, external rotation and internal rotation. The measured values are added to determine a combined value that is associated with a score from 0 to 5.
  * 211-300 degrees = 5 points
  * 161 to 210 degrees = 4 points
  * 101 to 160 degrees = 3 points
  * 61 to 100 degrees = 2 points
  * 31 to 60 degrees = 1 points
  * 0 to 30 degrees = 0 points
Time Frame: pre-operative, 1,3 and 5 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 221
Number analyzed (Hips) | 240
units on a scale
  HHS ROM Mean Preoperative Score | 3.90 (0.95)
  HHS ROM Mean 1 Year Score: number analyzed (Participants) | 194
  HHS ROM Mean 1 Year Score: number analyzed (Hips) | 211
  HHS ROM Mean 1 Year Score | 4.99 (0.12)
  HHS ROM Mean 3 Year Score: number analyzed (Participants) | 147
  HHS ROM Mean 3 Year Score: number analyzed (Hips) | 158
  HHS ROM Mean 3 Year Score | 4.99 (0.11)
  HHS ROM Mean 5 Year Score: number analyzed (Participants) | 115
  HHS ROM Mean 5 Year Score: number analyzed (Hips) | 122
  HHS ROM Mean 5 Year Score | 4.93 (0.31)
Statistical Analysis 1: Comparison: Trident® X3 Polyethylene Insert; Change in Harris Hip ROM score from pre-op to 1 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 2: Comparison: Trident® X3 Polyethylene Insert; Change in Harris Hip ROM score from pre-op to 3 years; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 3: Comparison: Trident® X3 Polyethylene Insert; Change in Harris Hip ROM score from pre-op to 5 years; Test type: Superiority or Other; p < 0.0001, Sign test

9. Secondary Outcome: Mean SF-12 Health Survey Score to Assess Change
Description: Change in the SF-12 score is reported by comparing the mean preoperative, 1,3 and 5 year postoperative scores.The SF-12 Health Survey is a 12-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: pre-operative, 1,3 and 5 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 215
Number analyzed (Hips) | 233
units on a scale
  Mean SF-12 Physical Score Preoperative | 32.11 (8.86)
  Mean SF-12 Physical Score 1 year: number analyzed (Participants) | 194
  Mean SF-12 Physical Score 1 year: number analyzed (Hips) | 211
  Mean SF-12 Physical Score 1 year | 49.90 (8.51)
  Mean SF-12 Physical Score 3 years: number analyzed (Participants) | 138
  Mean SF-12 Physical Score 3 years: number analyzed (Hips) | 149
  Mean SF-12 Physical Score 3 years | 49.97 (8.74)
  Mean SF-12 Physical Score 5 years: number analyzed (Participants) | 117
  Mean SF-12 Physical Score 5 years: number analyzed (Hips) | 126
  Mean SF-12 Physical Score 5 years | 49.08 (8.38)
  Mean SF-12 Mental Score Preoperative | 53.75 (10.91)
  Mean SF-12 Mental Score 1 year: number analyzed (Participants) | 194
  Mean SF-12 Mental Score 1 year: number analyzed (Hips) | 211
  Mean SF-12 Mental Score 1 year | 55.72 (7.83)
  Mean SF-12 Mental Score 3 years: number analyzed (Participants) | 138
  Mean SF-12 Mental Score 3 years: number analyzed (Hips) | 149
  Mean SF-12 Mental Score 3 years | 55.78 (8.13)
  Mean SF-12 Mental Score 5 years: number analyzed (Participants) | 117
  Mean SF-12 Mental Score 5 years: number analyzed (Hips) | 126
  Mean SF-12 Mental Score 5 years | 54.88 (7.76)
Statistical Analysis 1: Comparison: Trident® X3 Polyethylene Insert; Change in SF-12 Phyiscal Component Score from preop to 1 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 2: Comparison: Trident® X3 Polyethylene Insert; Change in SF-12 Phyiscal Component Score from preop to 3 year; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Trident® X3 Polyethylene Insert; Change in SF-12 Phyiscal Component Score from preop to 5 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 4: Comparison: Trident® X3 Polyethylene Insert; Change in SF-12 Mental Component Score from preop to 1 year; Test type: Superiority or Other; p = 0.0242, Sign test
Statistical Analysis 5: Comparison: Trident® X3 Polyethylene Insert; Change in SF-12 Mental Component Score from preop to 3 year; Test type: Superiority or Other; p = 0.0247, Sign test
Statistical Analysis 6: Comparison: Trident® X3 Polyethylene Insert; Change in SF-12 Mental Component Score from preop to 5 year; Test type: Superiority or Other; p = 0.1372, Sign test

10. Secondary Outcome: Mean Lower Extremity Activity Scale (LEAS) Score to Assess Change
Description: Change in the LEAS is reported by comparing the mean preoperative, 1,3 and 5 year scores. The LEAS is completed by the participant to assess activity level. Activity levels are ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: pre-operative, 1,3 and 5 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 221
Number analyzed (Hips) | 240
units on a scale
  Mean LEAS score Preoperative | 8.95 (2.54)
  Mean LEAS score 1 year: number analyzed (Participants) | 198
  Mean LEAS score 1 year: number analyzed (Hips) | 215
  Mean LEAS score 1 year | 11.65 (3.01)
  Mean LEAS score 3 years: number analyzed (Participants) | 141
  Mean LEAS score 3 years: number analyzed (Hips) | 152
  Mean LEAS score 3 years | 11.69 (2.95)
  Mean LEAS score 5 years: number analyzed (Participants) | 122
  Mean LEAS score 5 years: number analyzed (Hips) | 131
  Mean LEAS score 5 years | 10.92 (2.92)
Statistical Analysis 1: Comparison: Trident® X3 Polyethylene Insert; Change in LEAS Score from preop to 1 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 2: Comparison: Trident® X3 Polyethylene Insert; Change in LEAS Score from preop to 3 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 3: Comparison: Trident® X3 Polyethylene Insert; Change in LEAS Score from preop to 5 year; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

11. Secondary Outcome: Implant Survivorship
Description: Implant survivorship is determined using the Kaplan-Meier method.
Time Frame: 10 years
Population: Participants with available data. The population includes all 240 cases who were initially consented to 5 year study.
  There are 127 cases who consented to continue in the 10 year study.
Measure: Number; unit: percentage of hips
Units Other Than Participants: hips
Arm/Group | Trident® X3 Polyethylene Insert
Number analyzed (Participants) | 221
Number analyzed (hips) | 240
percentage of hips
  Kaplan-Meier Estimate (based on 5 year cases) | 95.79
  Kaplan-Meier Estimate (based on 10 year cases): number analyzed (Participants) | 116
  Kaplan-Meier Estimate (based on 10 year cases): number analyzed (hips) | 127
  Kaplan-Meier Estimate (based on 10 year cases) | 98.37

ADVERSE EVENTS:
Time Frame: To 10 yrs postop. Initially, all AEs reported then modified to operative-site (serious/non-serious) and serious systemic. Yrs 6-10 op-site (serious/non-serious) & any AE deemed to be related or uncertain in relation to device.
Description: Censored were not included as at risk. Industry Standard AE terms not used; specific AE terms not used for all AEs. Elective procedures not included eg. non-study joint replacement/revision, rotator cuff repair, carpal tunnel release, cataract, intra-ocular & bunion procedures, total shoulder repair, laminectomy, microdiscectomy, breast reduction, cervical spine fusion & mid-foot/flat-foot surgery.
Groups:
- Operative Adverse Events: Trident X3 Polyethylene Insert. Operative site events are reported by hip because in the case of bilateral participants (this is when one participant has both hips enrolled in the study), an event can occur in one hip, both hips or the same hip at different times and are counted separately for this reason.
- Non-operative Adverse Events: Trident X3 Polyethylene Insert. Non-operative site events are reported by participant.
Arm/Group | Operative Adverse Events | Non-operative Adverse Events
Serious Adverse Events (participants affected / at risk) | 12/240 | 33/221
Other Adverse Events (participants affected / at risk) | 62/240 | 65/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=240) | Non-operative Adverse Events (N=221)
Non-operative Site (Cardiac disorders) | 0/0 (0) | 3 (3)
Non-operative Site (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Non-operative Site (General disorders) | 0/0 (0) | 1 (1)
Non-operative Site (Hepatobiliary disorders) | 0/0 (0) | 1 (1)
Operative Site (Infections and infestations) | 1 (1) | 0/0 (0)
Non-operative Site (Infections and infestations) | 0/0 (0) | 4 (4)
Operative Site (Injury, poisoning and procedural complications) | 1 (1) | 0/0 (0)
Operative Site (Musculoskeletal and connective tissue disorders) | 11 (19) | 0/0 (0)
Non-operative Site (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 13 (14)
Non-operative Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 4 (4)
Operative Site (Nervous system disorders) | 1 (1) | 0/0 (0)
Non-operative Site (Nervous system disorders) | 0/0 (0) | 1 (1)
Non-operative Site (Psychiatric disorders) | 0/0 (0) | 1 (1)
Non-operative Site (Renal and urinary disorders) | 0/0 (0) | 3 (3)
Non-operative Site (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Non-operative Site (Vascular disorders) | 0/0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=240) | Non-operative Adverse Events (N=221)
Non-operative Site (Blood and lymphatic system disorders) | 0/0 (0) | 17 (17)
Non-operative Site (Infections and infestations) | 0/0 (0) | 13 (15)
Operative Site (Injury, poisoning and procedural complications) | 19 (19) | 0/0 (0)
Operative Site (Musculoskeletal and connective tissue disorders) | 45 (55) | 0/0 (0)
Non-operative Site (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 41 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study.These manuscripts and abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the sponsor for review at least 60 days prior to submission for publication.The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.